CLINICAL TRIAL: NCT01028703
Title: Does a Reduction in Renal Function Increase Arterial Stiffness and Left Ventricular Mass? - A Prospective Study of Kidney Donors
Brief Title: Effects of a Reduction in Kidney Function on Cardiovascular Structure and Function: A Prospective Study of Kidney Donors
Status: Completed | Type: Observational
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, William E Moody, BHF Clinical Research Fellow, University Hospital Birmingham NHS Foundation Trust
Other Study IDs: RKK3922
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic kidney disease; left ventricular dysfunction; diastolic dysfunction; hypertension
MeSH Terms: conditions — Renal Insufficiency, Chronic; Ventricular Dysfunction, Left; Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Donors: 110 will be "cases" that undergo uninephrectomy
- Controls: 110 "controls"

SUMMARY:
Studies of patients with established kidney disease, even when this is mild, appear to show that they are at high risk of heart failure, stroke and sudden cardiac death. This may be because kidney disease causes stiffening of the arteries in the body which means that the heart and brain are damaged by high blood pressure. By studying patients before and after the removal of a kidney (uni-nephrectomy) for transplantation the investigators will find out for the first time in man the effect of an isolated reduction in kidney function on the structure and function of the arteries and heart.

Hypotheses. An isolated reduction in GFR occuring after surgical uni-nephrectomy is associated with long term adverse cardiac and vascular effects which include:

1. Increased arterial stiffness and left ventricular mass
2. Abnormalities in left ventricular systolic and diastolic function
3. Increased oxidative stress, inflammation and collagen turnover

ELIGIBILITY:
Inclusion Criteria:

* Potential kidney donor attending University Hospital Birmingham NHS Foundation Trust

Current nationally set Exclusion Criteria:

* Diabetes mellitus
* Atrial fibrillation
* Left ventricular dysfunction (ejection fraction <40% on transthoracic echocardiography)
* History of cardiovascular or pulmonary disease
* Evidence of hypertensive end-organ damage.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Renal outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2010-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Left ventricular mass as measured by CMR and Echocardiography | 3 years
Arterial stiffness as measured by pulse wave velocity | 3 years

SECONDARY OUTCOMES:
Aortic compliance measured by cardiac magnetic resonance imaging | 3 years
Left ventricular systolic and diastolic elastance measured by echocardiography; | 3 years
Oxidative stress, inflammation and collagen turnover measured by blood assays of plasma renin, aldosterone, high sensitivity C-reactive protein (hsCRP), procollagen type III aminoterminal peptide (PIIINP) and C-telopeptide for type I collagen (CITP). | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan N Townend, Principal Investigator — Univeristy Hospital Birmingham NHS Foundation Trust
Locations (1):
- University Hospital Birmingham NHS Foundation Trust, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Derived] Moody WE, Ferro CJ, Edwards NC, Chue CD, Lin EL, Taylor RJ, Cockwell P, Steeds RP, Townend JN; CRIB-Donor Study Investigators. Cardiovascular Effects of Unilateral Nephrectomy in Living Kidney Donors. Hypertension. 2016 Feb;67(2):368-77. doi: 10.1161/HYPERTENSIONAHA.115.06608. PMID 26754643